CLINICAL TRIAL: NCT00144963
Title: Phase I-II Study of Liposomal Vincristine (VSLI) and Dexamethasone in Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Liposomal Vincristine Plus Dexamethasone in Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSLI-06-ALL
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VSLI (Experimental): Vincristine Sulfate Liposomes Injection (VSLI)
  Interventions: Drug: Vincristine Sulfate Liposomes Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vincristine Sulfate Liposomes Injection — Study treatment consists of infusion of VSLI intravenously over 60 minutes on Day 1 and Days 8, 15 and 22 (+/- 2 days).
  Other Names: Marqibo
Drug: Dexamethasone — Study treatment consists of 40 mg dexamethasone, daily orally or intravenously, on Days 1-4 (+/- 2 days) and Days 11-14 (+/- 2 days).

SUMMARY:
The purpose of this study is to find the highest safe dose and to assess the anti-tumor effect of liposomal vincristine with dexamethasone in patients with relapsed or refractory acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of liposomal vincristine given with dexamethasone in patients with relapsed or refractory acute lymphoblastic leukemia (ALL).
* Determine the efficacy of liposomal vincristine given with dexamethasone in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated, relapsed or refractory ALL (including lymphoblastic lymphoma and Burkitt's subtypes) with measurable disease.
* Performance status ≤3 (ECOG).
* All ages are eligible. Those aged 12 years or older may be counted towards the MTD in the Phase I portion of the trial. Pediatric patients are eligible, but must be treated at a dose level previously tested in an adult (one full course).
* Adequate liver function (bilirubin ≤2 x upper limit normal), and renal function (creatinine ≤2 x upper limit normal).
* Negative pregnancy test in females of childbearing potential.
* Patients with prior history of stem cell transplant are eligible if they meet all other eligibility requirements.

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics.
* Treatment with any investigational agents or chemotherapy agents in the last 21 days before study entry, unless full recovery from side effects has occurred or the patient has rapidly progressive disease judged to be life threatening by the Investigator.
* Concurrent treatment with other anti-cancer agents other than dexamethasone.
* Known CNS leukemia or lymphoma requiring intrathecal or craniospinal radiation therapy or with CNS neuropathy limiting evaluation of study drug. Patients with controlled CNS disease (no progression signs or symptoms at the time of study entry) may be eligible after approval by the Principal Investigator. Lumbar puncture not required in asymptomatic patients.
* Prior history of Grade 3 or 4 sensory or motor neuropathy related to chemotherapeutic treatment, or persistent Grade 2 or greater active neuropathy.
* History of active neurologic disorders unrelated to chemotherapy (including familial neurologic diseases and acquired demyelinating disorders).
* Prior history of hypersensitivity reactions to vincristine or any of the other components of VSLI.
* Pregnant and/or lactating women; or fertile men or women not willing to use contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Thomas, MD, Principal Investigator — MD Anderson Cancer Center, Department of Hematology/Oncology; Wendy Stock, MD, Principal Investigator — University of Chicago; Leonard Heffner, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VSLI
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VSLI
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: MTD of VSLI
Description: Subjects had to receive at least 1 course consisting of 4 weekly infusions of VSLI at the assigned drug dose with a minimum 2 weeks of observation after the last VSLI dose to be included in the evaluation of the MTD.
Time Frame: 6 weeks
Population: This study was designed to define the MTD of VSLI. Up to 7 sequential escalating dose cohorts (1.5, 1.825, 2.0, 2.25, 2.4, 2.6, and 2.8 mg/m2) were planned, with at least 3 subjects in each cohort. Escalation to the next higher dose cohort was allowed to proceed only if no nonhematologic DLT was observed.
Measure: Number; unit: mg/m2
Arm/Group | VSLI
Number analyzed (Participants) | 26
mg/m2 | 2.25

ADVERSE EVENTS:
Time Frame: start of dosing until 30 days after permanent discontinuation of study treatment or until permanent discontinuation of study treatment and initiation of a subsequent anti-leukemia therapy
Arm/Group | VSLI
Serious Adverse Events (participants affected / at risk) | 33/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VSLI (N=36)
Bacteraemia (Infections and infestations) | 17
Pneumonia, fungal (Infections and infestations) | 3
pneumonia (Infections and infestations) | 2
febrile neutropenia (Blood and lymphatic system disorders) | 12
neutropenia (Blood and lymphatic system disorders) | 3
pyrexia (General disorders) | 10
abdominal pain (Gastrointestinal disorders) | 4
oesophagitis (Gastrointestinal disorders) | 2
dehydration (Metabolism and nutrition disorders) | 3
failure to thrive (Metabolism and nutrition disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 2
hypotension (Vascular disorders) | 7
alanine aminotransferase increased (Investigations) | 2
aspartate aminotransferase increased (Investigations) | 2
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
peripheral neuropathy (Nervous system disorders) | 2
confusional state (Psychiatric disorders) | 2
mental status changes (Psychiatric disorders) | 2
cardiac arrest (Cardiac disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VSLI (N=36)
hyperglycaemia (Metabolism and nutrition disorders) | 15
hypokalaemia (Metabolism and nutrition disorders) | 10
decreased appetite (Metabolism and nutrition disorders) | 9
hypomagnesaemia (Metabolism and nutrition disorders) | 9
dehydration (Metabolism and nutrition disorders) | 8
hypocalcaemia (Metabolism and nutrition disorders) | 6
hyperphosphataemia (Metabolism and nutrition disorders) | 3
hyponatraemia (Metabolism and nutrition disorders) | 3
hypophosphataemia (Metabolism and nutrition disorders) | 3
failure to thrive (Metabolism and nutrition disorders) | 2
hyperkalaemia (Metabolism and nutrition disorders) | 2
hyperuricaemia (Metabolism and nutrition disorders) | 2
metabolic acidosis (Metabolism and nutrition disorders) | 2
anaemia (Blood and lymphatic system disorders) | 17
febrile neutropenia (Blood and lymphatic system disorders) | 14
neutropenia (Blood and lymphatic system disorders) | 13
thrombocytopenia (Blood and lymphatic system disorders) | 13
leukopenia (Blood and lymphatic system disorders) | 2
fatigue (General disorders) | 22
pyrexia (General disorders) | 18
chills (General disorders) | 12
oedema peripheral (General disorders) | 7
oedema (General disorders) | 5
asthenia (General disorders) | 4
chest pain (General disorders) | 4
pain (General disorders) | 2
neuropathy peripheral (Nervous system disorders) | 19
dizziness (Nervous system disorders) | 10
headache (Nervous system disorders) | 9
paraesthesia (Nervous system disorders) | 8
hypoaesthesia (Nervous system disorders) | 4
peripheral sensory neuropathy (Nervous system disorders) | 4
encephalopathy (Nervous system disorders) | 3
peripheral motor neuropathy (Nervous system disorders) | 3
dysgeusia (Nervous system disorders) | 2
neuralgia (Nervous system disorders) | 2
tremor (Nervous system disorders) | 2
constipation (Gastrointestinal disorders) | 24
nausea (Gastrointestinal disorders) | 17
abdominal pain (Gastrointestinal disorders) | 16
diarrhoea (Gastrointestinal disorders) | 15
abdominal distension (Gastrointestinal disorders) | 8
gatrooesophageal reflux disease (Gastrointestinal disorders) | 7
vomitting (Gastrointestinal disorders) | 6
abdominal discomfort (Gastrointestinal disorders) | 3
dyspepsia (Gastrointestinal disorders) | 3
dry mouth (Gastrointestinal disorders) | 2
gingival bleeding (Gastrointestinal disorders) | 2
oesophagitis (Gastrointestinal disorders) | 2
pancreatitis (Gastrointestinal disorders) | 2
rectal haemorrhage (Gastrointestinal disorders) | 2
myalgia (Musculoskeletal and connective tissue disorders) | 13
bone pain (Musculoskeletal and connective tissue disorders) | 12
arthralgia (Musculoskeletal and connective tissue disorders) | 6
muscular weakness (Musculoskeletal and connective tissue disorders) | 6
back pain (Musculoskeletal and connective tissue disorders) | 4
pain in extremity (Musculoskeletal and connective tissue disorders) | 4
muscle spasms (Musculoskeletal and connective tissue disorders) | 3
flank pain (Musculoskeletal and connective tissue disorders) | 2
myopathy (Musculoskeletal and connective tissue disorders) | 2
bacteraemia (Infections and infestations) | 9
staphylococcal bacteraemia (Infections and infestations) | 4
pneumonia (Infections and infestations) | 3
pneumonia fungal (Infections and infestations) | 3
bacterial infection (Infections and infestations) | 2
enterococcal bacteraemia (Infections and infestations) | 2
sepsis (Infections and infestations) | 2
urinary tract infection (Infections and infestations) | 2
alanine aminotransferase increased (Investigations) | 9
aspartate aminotransferase increased (Investigations) | 8
blood lactate dehydrogenase increased (Investigations) | 6
blood alkaline phosphatase increased (Investigations) | 4
blood urea increased (Investigations) | 4
cough (Respiratory, thoracic and mediastinal disorders) | 11
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
hiccups (Respiratory, thoracic and mediastinal disorders) | 5
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3
rhinitis alergic (Respiratory, thoracic and mediastinal disorders) | 3
atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
epistasis (Respiratory, thoracic and mediastinal disorders) | 2
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
insomnia (Psychiatric disorders) | 16
anxiety (Psychiatric disorders) | 7
confusional state (Psychiatric disorders) | 7
mental status change (Psychiatric disorders) | 4
depression (Psychiatric disorders) | 2
sleep disorder (Psychiatric disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 5
petechiae (Skin and subcutaneous tissue disorders) | 4
dry skin (Skin and subcutaneous tissue disorders) | 3
ecchymosis (Skin and subcutaneous tissue disorders) | 2
erythema (Skin and subcutaneous tissue disorders) | 2
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
night sweats (Skin and subcutaneous tissue disorders) | 2
hypotension (Vascular disorders) | 12
hypertension (Vascular disorders) | 5
tachycardia (Cardiac disorders) | 9
cardiac arrest (Cardiac disorders) | 2
sinus tachycardia (Cardiac disorders) | 2
vision blurred (Eye disorders) | 5
hyperbilirubinaemia (Hepatobiliary disorders) | 3
contusion (Injury, poisoning and procedural complications) | 3
vaginal haemorrhage (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less